CLINICAL TRIAL: NCT06304116
Title: Effect of Lidocaine Block in Traumatic Brain Injury: A Double-blind Randomized Controlled Study
Brief Title: Effect of Lidocaine Block in Traumatic Brain Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad (Other)
Responsible Party: Sponsor-Investigator, Muhammad, Research Director, Ahmadu Bello University Teaching Hospital
Organization: Ahmadu Bello University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGB-TBI
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Rehabilitation; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation therapy+Stellate ganglion block (Experimental): The study lasted 10 days for each patient. During the treatment, All the participants were provided with the rehabilitation therapy, which included routine rehabilitation, cognitive training, swallowing function training and nutrition support.
  Based on the invention above, the patients in the observation group were provided with stellate ganglion block, using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g)
  Interventions: Behavioral: Rehabilitation therapy; Procedure: Stellate ganglion block; Drug: Lidocaine Hydrochloride
- Rehabilitation therapy+Placebo (Placebo Comparator): The study lasted 10 days for each patient. During the treatment, All the participants were provided with the rehabilitation therapy, which included routine rehabilitation, cognitive training, swallowing function training and nutrition support.
  Interventions: Behavioral: Rehabilitation therapy; Procedure: Stellate ganglion block

INTERVENTIONS:
Behavioral: Rehabilitation therapy — During the treatment, All the participants were provided with the rehabilitation therapy, which included routine rehabilitation, cognitive training, swallowing function training and nutrition support.
Procedure: Stellate ganglion block — The percutaneous approach via the paratracheal route was used for Stellate ganglion block . The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
Drug: Lidocaine Hydrochloride — Based on the invention above, the patients in the observation group were provided with Stellate ganglion block , using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g). The percutaneous approach via the paratracheal route was used for Stellate ganglion block . The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Arms: Rehabilitation therapy+Stellate ganglion block

SUMMARY:
The goal of this or clinical trial is to explore efficacy of stellate ganglion block on dysphagia and activities of daily living in Traumatic Brain Injury Patients. The main question it aims to answer are:

Can stellate ganglion block improve the dysphagia and activities of daily living in Traumatic Brain Injury Patients.

Traumatic Brain Injury Patients will be divided into the the control group and observation group evenly. All the patients were provided with routine therapy, while the patients in the observation group were given stellate ganglion block. The swallowing function, and activities of daily living of the two groups of patients before and after treatment were evaluated.

DETAILED DESCRIPTION:
Dysphagia, or swallowing difficulty, is a common symptom in Traumatic Brain Injury Patients. The goal of this or clinical trial is to explore efficacy of stellate ganglion block on dysphagia and activities of daily living in Traumatic Brain Injury Patients. The main question it aims to answer are:

Can stellate ganglion block improve the dysphagia and activities of daily living in Traumatic Brain Injury Patients.

Traumatic Brain Injury Patients will be divided into the the control group and observation group evenly. All the patients were provided with routine therapy, while the patients in the observation group were given stellate ganglion block. The swallowing function, and activities of daily living of the two groups of patients before and after treatment were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years, meeting the diagnosis of Traumatic Brain Injury;
* presence of no contraindication for Stellate Ganglion Block;
* with stable vital signs and no severe liver or kidney dysfunction, metabolic disorders.
* informed consent form was obtained from the patient's family members, indicating their full - understanding of the study and agreement to participate.

Exclusion Criteria:

* unable to cooperate in completing treatment and assessment due to personal reasons or other disorders;
* complicated with other intracranial lesions, such as stroke;
* with severe consciousness disorders caused by other diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale | day 1 and day 10
  Penetration-Aspiration Scale is used to assess dysphagia under Videofluoroscopic Swallowing Study, primarily evaluating the extent to which fluid food enter the airway and caused penetration or aspiration during the swallowing process. As the level increases, the severity of dysphagia also increases. The score ranges 1 to 8.

SECONDARY OUTCOMES:
Modified Barthel Index | day 1 and day 10
  The activities of daily living of patients will be assessed using the modified Barthel Index . The scale includes 10 items such as feeding, bathing, walking, dressing. Each item is rated on a 4-point scale based on the level of assistance required, with a total score of 100 points. There is a positive correlation between activities of daily living and the final score.The score ranges 1 to 100.
Swallowing duration | day 1 and day 10
  The time duration that the patient swallowed the contrast agent under Videofluoroscopic Swallowing Study the is recorded.Unit: seconds.
Functional Oral Intake Scale | day 1 and day 10
  During Dysphagia-Functional Oral Intake Scale assessment, evaluators engage in communication with the patient, conduct observations, and make records to assess the patient's oral intake ability. The Functional Oral Intake Scale assessment form includes seven levels of scoring, ranging from level 1 to level 7, indicating a progressive improvement in the patient's oral intake ability.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Director — Site Coordinator of United Medical Group